CLINICAL TRIAL: NCT01314742
Title: A Randomized Controlled Clinical Trial of Two Different Oral Care Regimens Combined With Ventilator-Associated Pneumonia (VAP) Bundle Strategy for Reduction of Duration of Mechanical Ventilation in a Neonatal Population
Brief Title: Study of Biotene OralBalance Gel for Oral Care in Critically-Ill Mechanically Ventilated Neonates
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00013036; FMC 2010-100 (Other: Forsyth Medical Center IRB)
Record Dates: First submitted 2011-03-09; First posted 2011-03-14 (Estimated); Results first posted 2014-02-04 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Ventilator-associated Pneumonia
Keywords: neonates; mechanical ventilation; oral care; duration of mechanical ventilation; feasibility; ventilator-associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biotene OralBalance® gel Arm (Experimental): Biotene OralBalance® gel contains antibacterial active ingredients: lactoperoxidase, lysozyme and lactoferrin. These enzymes occur naturally in the human milk and colostrum and have mimicking properties of the human saliva activity in vivo.
  Interventions: Drug: Biotene OralBalance® gel
- Sterile Water Arm (Placebo Comparator): Sterile Water moisten cotton tipped applicator
  Interventions: Other: Sterile Water moisten cotton tipped applicator

INTERVENTIONS:
Drug: Biotene OralBalance® gel — Biotene OralBalance® gel is dispensed as 42gm, patient specific tube from hospital's Central Pharmacy. One pea-size oral application every 4 hours, or at touch time, to gums and tongue, as long as the subject remains mechanically ventilated for the duration of hospitalization.
  Arms: Biotene OralBalance® gel Arm
Other: Sterile Water moisten cotton tipped applicator — One oral care application will be performed every 4 hours, or at touch times, to gums and tongue, as long as the subject remains mechanically ventilated for the duration of hospitalization.
  Arms: Sterile Water Arm

SUMMARY:
The goal of this pilot study is to test the hypothesis that mechanically ventilated infants receiving Biotene OralBalance® gel for oral care would have a reduced intubation time compared to infants receiving oral care placebo. This study is also performed to test the feasibility as well the safety of Biotene OralBalance® gel.

DETAILED DESCRIPTION:
Prolonged mechanical ventilation is a known risk factor strongly associated with ventilator-associated pneumonia (VAP). As the fatality rates for VAP are high, prevention of VAP has focused on the use of "VAP bundles". Oral decontamination, by reducing the microbial burden within a patient's oral cavity, is an essential part of VAP bundle strategy for reducing VAP rates in mechanically ventilated adults and older children. However there are no published studies of oral care products for VAP prevention in mechanically ventilated neonates. Biotene OralBalance® gel contains antibacterial active ingredients, including lactoperoxidase, lysozyme and lactoferrin,all enzymes with bacteriostatic or bactericidal activity on selective oral microflora. We hypothesize that by directly reducing the oral microbial burden, we indirectly reduce the number of VAP. This will be reflected in the reduced time on mechanical ventilation in the group of infants receiving Biotene OralBalance® gel.

This is a prospective, randomized, unmasked, controlled trial with 40 mechanically ventilated infants recruited from level IV nursery at Forsyth Medical Center, Winston-Salem, NC. The participants will be randomized to two equal groups, stratified by gestational age categories: <28 weeks, and >=28 weeks as well as multiple births. Twenty infants will receive Biotene OralBalance® gel (Intervention Group) and 20 infants will receive swabs with sterile water (Control Group) for timed oral care. Both study groups will receive the NICU standard ventilator-associated pneumonia (VAP) bundle, a combination of strategies aimed to reduce the rate of VAP.

ELIGIBILITY:
Inclusion Criteria:

* Neonates who are mechanically ventilated between 7 and 10 days old. Signed parental informed consent is required for recruitment into the study.

Exclusion Criteria:

* Neonates with chromosomal anomalies or major congenital anomalies, neonates with terminal conditions, neonates for whom a decision has been made not to provide full medical support, neonates whose parents refused or are unable to provide consent, and/or attending physician refusal.

Min Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Stefanescu, MD, MS, Principal Investigator — Wake Forest University
Locations (2):
- United States (2):
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Brenner Children's Hospital, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tenovuo J. Clinical applications of antimicrobial host proteins lactoperoxidase, lysozyme and lactoferrin in xerostomia: efficacy and safety. Oral Dis. 2002 Jan;8(1):23-9. doi: 10.1034/j.1601-0825.2002.1o781.x. PMID 11936452
- [Background] Tenovuo J, Lumikari M, Soukka T. Salivary lysozyme, lactoferrin and peroxidases: antibacterial effects on cariogenic bacteria and clinical applications in preventive dentistry. Proc Finn Dent Soc. 1991;87(2):197-208. PMID 1896432
- [Background] Epstein JB, Emerton S, Le ND, Stevenson-Moore P. A double-blind crossover trial of Oral Balance gel and Biotene toothpaste versus placebo in patients with xerostomia following radiation therapy. Oral Oncol. 1999 Mar;35(2):132-7. doi: 10.1016/s1368-8375(98)00109-2. PMID 10435146
- [Background] Apisarnthanarak A, Holzmann-Pazgal G, Hamvas A, Olsen MA, Fraser VJ. Ventilator-associated pneumonia in extremely preterm neonates in a neonatal intensive care unit: characteristics, risk factors, and outcomes. Pediatrics. 2003 Dec;112(6 Pt 1):1283-9. doi: 10.1542/peds.112.6.1283. PMID 14654598
- [Background] Chlebicki MP, Safdar N. Topical chlorhexidine for prevention of ventilator-associated pneumonia: a meta-analysis. Crit Care Med. 2007 Feb;35(2):595-602. doi: 10.1097/01.CCM.0000253395.70708.AC. PMID 17205028
- [Result] Stefanescu BM, Hetu C, Slaughter JC, O'Shea TM, Shetty AK. A pilot study of Biotene OralBalance(R) gel for oral care in mechanically ventilated preterm neonates. Contemp Clin Trials. 2013 Jul;35(2):33-9. doi: 10.1016/j.cct.2013.03.010. Epub 2013 Apr 20. PMID 23608625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 82 mechanically ventilated infants ≤ 28 weeks gestation who were screened, 46 met eligibility criteria. Of these eligible infants 41(89%) were recruited and randomized.
Groups:
- Biotene OralBalance® Gel Arm: Biotene OralBalance® gel contains antibacterial active ingredients: lactoperoxidase, lysozyme and lactoferrin. These enzymes occur naturally in the human milk and colostrum and have mimicking properties of the human saliva activity in vivo.
  Biotene OralBalance® gel : Biotene OralBalance® gel is dispensed as 42gm, patient specific tube from hospital's Central Pharmacy. One pea-size oral application every 4 hours, or at touch time, to gums and tongue, as long as the subject remains mechanically ventilated for the duration of hospitalization.
- Sterile Water Arm: Sterile Water moisten cotton tipped applicator : One oral care application will be performed every 4 hours, or at touch times, to gums and tongue, as long as the subject remains mechanically ventilated for the duration of hospitalization.
Period: Overall Study
Arm/Group | Biotene OralBalance® Gel Arm | Sterile Water Arm
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biotene OralBalance® Gel Arm | Sterile Water Arm | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 21 | 41
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: gestational age (weeks)] | 24 (0) [24 to 25] | 25 (0) [24 to 25] | 24 (0) [24 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Description: percentage of participants with retention
Time Frame: duration of study, for up to 30 months
Measure: Number; unit: percentage of participants retained
Groups:
- Biotene OralBalance® Gel Arm: Study group receiving timed oral care with Biotene OralBalance® gel Arm
- Sterile Water Group: Study group receiving timed oral care with Sterile Water
Arm/Group | Biotene OralBalance® Gel Arm | Sterile Water Group
Number analyzed (Participants) | 20 | 21
percentage of participants retained | 100 | 100

2. Primary Outcome: Duration of Mechanical Ventilation
Description: Time on invasive mechanical ventilation will be measured in days
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: ventilator-days
Arm/Group | Biotene OralBalance® Gel Arm | Sterile Water Arm
Number analyzed (Participants) | 20 | 21
ventilator-days | 32 (15) | 30 (13)

ADVERSE EVENTS:
Time Frame: duration of intervention, for up to 30 months
Arm/Group | Biotene OralBalance® Gel Arm | Sterile Water Arm
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No